CLINICAL TRIAL: NCT03144570
Title: EURopean Study on Encephalitis in Intensive CAre
Acronym: EURECA
Status: Completed | Type: Observational
Sponsor: ICUREsearch (Industry)
Responsible Party: Sponsor
Other Study IDs: 0008
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Encephalitis
Keywords: ICU, encephalitis, meningo-encephalitis, seizures
MeSH Terms: conditions — Encephalitis; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None, non-interventional study — Not applicable, non-interventional study

SUMMARY:
Prospective observational multicenter study in European ICUs. All patients admitted to the ICU for probable or confirmed Acute encephalitis (2013 IDSA - Infectious Disease Society of America criteria) will be included. Factors associated with a poor prognosis will be identified by multivariate analysis using a logistic regression.

DETAILED DESCRIPTION:
Primary objective :

evaluate the correlation between mRs score and the baseline characteristics Functional outcomes will be evaluated using the modified Rankin score (mRS) score, which is one of the most frequently used scores in acute neurological diseases [18]. A poor outcome will be defined by a mRS score > 2 (functional dependence or death). The investigator usually evaluates this score if the patient is still in the hospital 90 days after admission. Patients discharged from hospital within 90 days following ICU admission without major disability (mRS 0, 1 or 2) are considered to have a good outcome. Patients discharged within 90 days with a disability will be classified for the study according to the latest available data. Patients will not be contacted directly by the investigator for the study purposes.

Secondary objectives :

To identify additional prognosis factors : the clinical, radiological, biological and neurophysiological factors associated with poor outcome for patients admitted to the ICU with AE

* Day 28 mortality, in-ICU mortality, in-hospital mortality
* Major systemic complications (septic shock, hyponatremia, nosocomial pneumonia, catheter-related BSI, overt gastroenteral bleeding, pulmonary embolism)
* Major intracranial complications during ICU stay

  * Status epilepticus
  * Brain death
  * Empyema/cerebral abscess
  * Cerebral ischemia
  * Intracranial bleeding
* ICP monitoring
* Neurosurgery

The cause of death will be categorized into 2 categories:

* Systemic causes (cardiovascular failure, MOF)
* Neurological cause (Diffuse neurologic injury or withdrawal of care)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* non-opposition to participate in the study (or consent if applicable according to local legislation)
* Impaired consciousness (altered mentation, stupor, or personality changes) for a duration ≥ 24 h, without obvious explanation
* A score on the Glasgow Coma Scale < or =13 at ICU admission
* A Cerebrospinal fluid pleocytosis > = 5 cell / mm3
* At least 2 of the following :

  * Fever (≥ 38.0 °C) within 72 hours before or after admission
  * Generalized or partial seizures non-attributable to pre-existing epilepsy
  * New onset focal neurological deficit
  * Parenchymal abnormalities on MRI compatible with AE
  * EEG alterations compatible with AE.

Exclusion Criteria:

* CSF or neuroimaging not available (s) or not performed.
* febrile encephalopathy associated with another diagnosis (sepsis, neurological disease with aspiration pneumonia ... )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 patients admitted to the ICU for AE (5 consecutive patients in each participating ICU, targeted number of ICUs in Europe : 200).
Sampling Method: Non-Probability Sample
Enrollment: 596 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Modified Rankin scale score | Day 90
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It has become the most widely used clinical outcome measure for stroke clinical trials.

SECONDARY OUTCOMES:
Mortality at Day 28 | Day 28
  Rate of death at day 28
Systematic complications | Day 90
  Septic shock, hyponatremia
Intracranial complications | Day 90
  Documented seizures, status epilepticus, Diffuse cerebral edema, herniation, Ischemia, cerebral hemorrhage
Intracranial pressure monitoring | Day 90
  List of all available methods of intracranial pressure monitoring used in study sites and their outcome
Neurosurgery | Day 90
  Monitoring of neurosurgery to identify additional prognosis factors

CONTACTS AND LOCATIONS:
Overall Officials: Jean François Timsit, Study Chair — ICUREsearch; Romain Sonneville, Principal Investigator — Hôpital Bichat, APHP
Locations (65):
- Medical University of Innsbruck, Innsbruck, Austria
- France (49):
  - Centre Hospitalier d'Angoulême, Angoulême
  - Centre Hospitalier Annecy Genevois, Annecy
  - Hôpital Victor Dupouy, Argenteuil
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU Brest, Brest
  - Hôpital Pierre Wertheimer, Bron
  - Centre Hospitalier René Dubos, Cergy-Pontoise
  - CH de Charlesville-Mézières, Charleville-Mézières
  - Les Hôpitaux de Chartres, Chartres
  - Centre Hospitalier Châlons en Champagne, Châlons-en-Champagne
  - Centre Hospitalier Public du Cotentin, Cherbourg
  - Hôpital Antoine Béclère, Clamart
  - CHU Gabriel Montpied, Clermont-Ferrand
  - APHP Colombes - Louis Mourier, Colombes
  - Centre Hospitalier du Sud Francilien, Corbeil-Essonnes
  - Hôpitaux Universitaires Henri Mondor, Créteil
  - Centre hopsitalier de Dieppe, Dieppe
  - Centre hospitalier Sud Essone, Étampes
  - CHU Grenoble, Grenoble
  - Marne la Vallée - Meaux, Jossigny
  - CH Vendée, La Roche
  - CH du Mans, Le Mans
  - Hôpital R Salengro, Lille
  - Centre Hospitalier Lorient, Lorient
  - Hôpital Edouard Herriot, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hôpital de la Timone, Marseille
  - CHU Hôpital Nord, Marseille
  - CHR Metz-Thionville, Metz
  - CHU Lapeyronie, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital de la Source, Orléans
  - Hôpital Saint Louis, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges-Pompidou, Paris
  - Hôpital Bichat Claude Bernard, Paris
  - Hôpitaux universitaires Est Parisien, Tenon, Paris
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Groupe hospitalier Pitié-Salpêtrière, Paris
  - Fondation Opthalmologique Adolphe de Rothschild, Paris
  - Centre Hospitalier de Pau, Pau
  - Centre Hospitalier Intercommunal de Poissy, Poissy
  - CHU Rennes, Rennes
  - CH Roanne, Roanne
  - Centre hospitalier de Saint-Denis, Hôpital DELAFONTAINE, Saint-Denis
  - CHU de Toulouse Purpan, Toulouse
  - Centre hospitalier de Tourcoing, Tourcoing
  - Hôpital André Mignot, Versailles
  - CH des 2 vallées, Site Longjumeau, Longjumeau, Île-de-France Region
- India (5):
  - Ims & Sum Hospital, Bhubaneswar
  - Sanjay Gandhi Post Graduate Institute of Medical Sciences, Lucknow
  - Institute Of Medical Sciences Banaras Hindu University, Lucknow
  - King George's medical university, Lucknow
  - Sri Ramachandra Institute of Higher Education and Research, Lucknow
- Italy (3):
  - Azienda USL Toscana Centro, Florence
  - San Gerardo Hospital, Monza
  - Università Cattolica del Sacro Cuore, Roma
- Academic Medical Center, Amsterdam, Netherlands
- Spain (6):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu, Barcelona
  - Germans Trias i Pujol, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitari Arnau de Vilanova, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonneville R, de Montmollin E, Contou D, Ferrer R, Gurjar M, Klouche K, Sarton B, Demeret S, Bailly P, da Silva D, Escudier E, Le Guennec L, Chabanne R, Argaud L, Ben Hadj Salem O, Thyrault M, Frerou A, Louis G, De Pascale G, Horn J, Helbok R, Geri G, Bruneel F, Martin-Loeches I, Taccone FS, De Waele JJ, Ruckly S, Staiquly Q, Citerio G, Timsit JF; EURECA Investigator Study Group. Clinical features, etiologies, and outcomes in adult patients with meningoencephalitis requiring intensive care (EURECA): an international prospective multicenter cohort study. Intensive Care Med. 2023 May;49(5):517-529. doi: 10.1007/s00134-023-07032-9. Epub 2023 Apr 6. PMID 37022378